CLINICAL TRIAL: NCT00646347
Title: A Pilot Study of Neuro Hand Orthosis Program: A Promising Restorative Therapy Treatment for the Severe Paralytic Arm in Subacute Stroke Rehabilitation
Brief Title: A Pilot Study of Neuro Hand Orthosis Program In Stroke Upper Limb Rehabilitation
Acronym: NHOP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St Luke's Hospital, Singapore (Other)
Collaborators: National Council Of Social Service, Singapore (Other)
Responsible Party: Gribson Chan Yu Chun Senior Rehabilitation Manager, St Luke's Hosptial
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: slhdoc02
Record Dates: First submitted 2008-03-24; First posted 2008-03-28 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2009-02

CONDITIONS: Paralytic Stroke
Keywords: stroke; upper limb rehabilitation; treatment; movement recovery from sever paralytic upper limb; neuro hand orthosis; self practice program; subacute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Conventional stroke upper limb rehabilitation is given
  Interventions: Other: Conventional upper limb stroke rehabilitation
- B (Active Comparator): Neuro Hand Orthosis Program is given
  Interventions: Device: Neuro Hand Orthosis Program (NHOP)

INTERVENTIONS:
Other: Conventional upper limb stroke rehabilitation — Patient will be given a ten weeks conventional upper limb therapy. 3 sessions will be provided weekly in the first 4 weeks and 2 therapy sessions will be provided weekly in the subsequent 6 weeks. Patients will receive half an hour of conventional therapy in each session.
  Patient will be taught to carry out two and half hours conventional self practice exercise daily for a period of ten weeks.
  Arms: A
Device: Neuro Hand Orthosis Program (NHOP) — The NHO is based on a design of dynamic hand orthosis for orthopaedic patients after hand surgery. We use it to support CVA patient's wrist and finger to perform grasping to transport an object (ball) from place to place to achieve the follows;
  1. NHO can assist stroke patients to experience successful hand grasping with an object and produce voluntary movement from their paralytic arm. This successful experience will positively reinforce the patient to continue to use their paralytic arm and change the patient's behavior and perception in the arm usage.
  2. The NHO Program is able to engage patients to perform their exercises and activities by themselves independently with the effect of intensive therapy.
  The intervention (NHOP) group will receive same treatment intensity as the control group but with a "Neuro Hand Orthosis".
  Arms: B

SUMMARY:
The implementation of Neuro Hand Orthosis Upper Limb Program can significantly improve the severe stroke paralytic arm in subacute rehabilitation as compared with the use of conventional therapy.

DETAILED DESCRIPTION:
The neuro hand orthosis is based on a design of dynamic hand orthosis for orthopaedic patients. We attempt to apply such an orthosis on stroke patients to aid in regaining movement from severe paralytic arm by helping the patients to support their wrist and finger in a functional position for grasping. The patient is then encouraged to produce voluntary movement from the severe paralytic arm to transport an object (ball) from place to place either in sitting or standing position.

Since intensive arm usage is associated with neuro reorganisation, we propose designing a program with the neuro hand to encourage usage of the paralysed hand and help overcome the barriers of poor motivation and lack of arm usage through self practice program.

ELIGIBILITY:
Inclusion Criteria:

* Post stroke between one week to three months and medically stable
* Right Hemiplegia with right hand dominant
* Able to stand with minimum assistance
* AMT score not lesser then 7/10
* Motricity Index Arm Score <36/100

Exclusion Criteria:

* Unable to commit to the Neuro Hand Orthosis Program (either as in or out patients) for 10 weeks according to the program regime or unable to follow the control group regime for 10 weeks
* Pre-existence shoulder or upper limb pain
* Pre-existence moderate or severe hand oedema
* Patients with terminal disease
* Resident of Institution (eg, Nursing home etc prior to admission)
* Pre-existing upper limb disability on affected arm
* Psychiatric problem

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-01 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Action Research Arm Test (ARAT) | week 4 , week 10 , 6 months and 12 months
Motricity Index | week 4 , week 10 , 6 months and 12 months

SECONDARY OUTCOMES:
Motor Activity Log (MAL) | At admission, week 4 , week 10 , 6 months and 12 months
Modified Ashworth Scale for grading Spasticity | At admission, week 4 , week 10 , 6 months and 12 months
Shoulder pain at admission | At admission, week 4 , week 10 , 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gribson Yu Chun Chan, Master, Principal Investigator — St Luke's Hospital, Singapore
Locations (1):
- St Luke's Hospital (Singapore), Singapore, 2 Bukit Batok, Street11, Singapore